CLINICAL TRIAL: NCT02986061
Title: To Catheterize or Not? in Total Knee Arthroplasty With Combined Spinal-epidural Analgesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Liu Yang, Director, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Knee-UC
Record Dates: First submitted 2016-11-30; First posted 2016-12-08 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Urinary Catheter
MeSH Terms: interventions — Urinary Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Active Comparator): Patients with indwelling urinary catheter
  Interventions: Device: Urinary catheter
- Study Group (No Intervention): Patients without indwelling urinary catheter

INTERVENTIONS:
Device: Urinary catheter
  Arms: Control Group

SUMMARY:
The aim of this study was to investigate whether urinary catheterization could be avoided for all patients undergoing total knee arthroplasty under combined spinal-epidural analgesia plus multi-site infiltration analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 years and older, who were scheduled for a primary TKA for end-stage osteoarthritis and those who were willing and able to return for follow-up over at least a 1-month postoperative period.

Exclusion Criteria:

* Revisions, bilateral procedures, surgical history of urinary system, urinary tract infection and systematical conditions (renal disease, renal failure, chronic renal insufficiency, or an indwelling catheter at the time of surgery) needing intraoperative monitoring urine output.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative urinary retention | 7 days
Postoperative urinary tract infection | 7 days
Urine volume | 3 days

SECONDARY OUTCOMES:
Length of stay | 14 days
Intraoperative intravenous fluid | 1 day
Duration of the surgery | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Joint Surgery, Southwest Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No